CLINICAL TRIAL: NCT03205566
Title: The Time to Protection and Adherence Requirements of Raltegravir With or Without Lamivudine in Protection From HIV Infection
Brief Title: Time to Protection and Adherence Requirements of Raltegravir With or Without Lamivudine in Protection From HIV Infection
Acronym: R-PrEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 202316
Record Dates: First submitted 2017-06-08; First posted 2017-07-02 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium; Lamivudine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A Raltegravir, then Raltegravir/Lamivudine (Active Comparator): 7 days Raltegravir 400mg bd followed by minimum 4 weeks wash out and then 7 days Raltegravir 400mg/lamivudine 150mg (oral tablets) bd.
  Interventions: Drug: Raltegravir 400Mg Tab; Drug: Lamivudine 150Mg Tablet
- Arm B Raltegravir/Lamivudine, then Raltegravir (Active Comparator): Raltegravir 400mg + Lamivudine 150mg tablet, taken twice a day for 7days followed by a minimum of 4 weeks wash out and then 7 days Raltegravir 400mg bd.
  Interventions: Drug: Raltegravir 400Mg Tab; Drug: Lamivudine 150Mg Tablet

INTERVENTIONS:
Drug: Raltegravir 400Mg Tab — bd for 7 days
  Other Names: Isentress
Drug: Lamivudine 150Mg Tablet — + Raltegravir 400Mg tablet bd for 7 days
  Other Names: Epivir

SUMMARY:
This study evaluates whether a 7-day course of Raltegravir 400mg bd or Raltegravir 400mg/lamivudine 150mg bd can prevent HIV from infecting genital tissue and will relate the level of drug in the blood to the level of drug in genital tissue and to the ability to of HIV to infect genital tissue. As well as determining whether these regimes can provide ex vivo protection against HIV, this study will also determine speed to provision of protection and a 48 hour PK/PD decay profile of Raltegravir following drug cessation after attaining steady state concentrations. The results will also inform all future HIV pre-exposure prophylaxis studies of Raltegravir and form the basis for large scale clinical trials without the need for tissue sampling. To date, efficacy studies assessing PrEP regimens have utilized HIV-acquisition endpoints with the consequence being such studies are required to be large in subject number in order to power observations. In addition the study will provide for the first time data on HIV protection rather than just Raltegravir drug levels in tissue, and allow assessment of the possibility of Raltegravir being used as an intermittent dosing regimen in PrEP.

DETAILED DESCRIPTION:
This is a multi-site, open-label, randomised, pharmacokinetic (PK) and pharmacodynamic (PD) trial whereby 36 individuals (18 women and 18 men) will be randomised according to gender 1:1:1:1:1:1 to one of 6 arms (A 1 A 2 A 3 B 1 B 2 B 3). The result being 3 women and 3 men will be in each arm. The letter dictates the ART regimen order and the number dictates the time points that tissue sampling will occur on and off ART. Two ART regimes will be investigated and all individuals will receive both regimes separated by a one month wash out.

Arm A (A 1 A 2 A 3): will start with 7 days Raltegravir 400mg bd and then have a one month wash out before then starting 7 days Raltegravir 400mg /lamivudine 150mg bd.

Arm B (B 1 B 2 B 3): will start with 7 days Raltegravir 400mg /lamivudine 150mg bd and then have a one month wash out before then starting 7 days Raltegravir 400mg bd. This will remove sequential selection bias. All individuals will receive tissue sampling at baseline for ex vivo analysis to ensure biopsies are infectable on challenge assays. Sampling from women will avoid menstruation and if possible focus on the luteal phase of the menstrual cycle. Individuals will receive another set of tissue sampling during and after ART in phase 1, have a 4 week wash out period and then have another set of sampling during and after ART in phase 2. Individuals will therefore have 5 sets of sampling during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and sign a written informed consent form prior to participation in any screening procedures and must be willing to comply with all trial requirements.
2. Male or non-pregnant, non-lactating females
3. Age between 18 to 60 years, inclusive.
4. Body Mass Index (BMI) of 16 to 35 kg/m2, inclusive.
5. Negative antibody/antigen combined test for HIV.
6. Absence of any significant health problems (in the opinion of the investigator) on the basis of the screening procedures; including medical history, physical examination, vital signs.
7. Women participating in sexual intercourse that could result in pregnancy -must use an adequate form of contraception throughout the study and for two weeks after the study. This includes intrauterine device, condoms, anatomical sterility in self or partner. Oral hormonal methods and implant contraceptives are allowed but only in combination with the additional protection of a barrier method.
8. Female participants may not use any vaginal products or objects or have vaginal sex for 48 hours before and after the collection of vaginal fluid and vaginal biopsies. This list includes tampons, female condoms, cotton wool, rags, diaphragms, cervical caps (or any other vaginal barrier method),douches, lubricants, vibrators/dildos, and drying agents.
9. Males participating in sexual intercourse that could result in pregnancy must use condoms during the duration of the study.
10. Men and women cannot use anal products or objects including but not exclusive to douches, lubricants and vibrators/dildos, butt plugs or urethral sounds or have receptive anal intercourse for 48 hours before and after the collection of rectal biopsies.
11. Willing to abstain from multivitamins and antacids for the study duration.

Exclusion Criteria:

1. Any significant acute or chronic medical illness.
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs or clinical laboratory determinations.
3. Positive blood screen for syphilis, hepatitis B (HBs Ag) and/or C antibodies.
4. Positive blood screen for HIV antibodies.
5. Positive screen for sexually transmitted infections at screening visit
6. High-risk behaviour for HIV infection which is defined as having one of the following within three months before trial day 0 (first dose): had unprotected vaginal or anal sex with a known HIV infected person or a casual partner. engaged in sex work for money or drugs. acquired a bacterial sexually transmitted disease in the past 3 months. having a known HIV positive partner either currently or in the previous six months Females who are pregnant or breast-feeding.
7. Clinically significant laboratory abnormalities (according to normal range as defined by central laboratory).
8. Participation in a clinical trial of an Investigational product within 1 month of planned baseline enrolment in this study.
9. Ingestion of H2 receptor antagonists or proton pump inhibitor drugs in the preceding 14 days
10. Current of planned use of anti-epileptics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Fox, Study Director — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Harrison Wing, Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Background] Garcia-Lerma JG, Otten RA, Qari SH, Jackson E, Cong ME, Masciotra S, Luo W, Kim C, Adams DR, Monsour M, Lipscomb J, Johnson JA, Delinsky D, Schinazi RF, Janssen R, Folks TM, Heneine W. Prevention of rectal SHIV transmission in macaques by daily or intermittent prophylaxis with emtricitabine and tenofovir. PLoS Med. 2008 Feb;5(2):e28. doi: 10.1371/journal.pmed.0050028. PMID 18254653
- [Background] Herrera C, Cranage M, McGowan I, Anton P, Shattock RJ. Colorectal microbicide design: triple combinations of reverse transcriptase inhibitors are optimal against HIV-1 in tissue explants. AIDS. 2011 Oct 23;25(16):1971-9. doi: 10.1097/QAD.0b013e32834b3629. PMID 21811139
- [Background] Anton PA, Saunders T, Elliott J, Khanukhova E, Dennis R, Adler A, Cortina G, Tanner K, Boscardin J, Cumberland WG, Zhou Y, Ventuneac A, Carballo-Dieguez A, Rabe L, McCormick T, Gabelnick H, Mauck C, McGowan I. First phase 1 double-blind, placebo-controlled, randomized rectal microbicide trial using UC781 gel with a novel index of ex vivo efficacy. PLoS One. 2011;6(9):e23243. doi: 10.1371/journal.pone.0023243. Epub 2011 Sep 28. PMID 21969851
- [Background] O'Quigley J, Zohar S. Experimental designs for phase I and phase I/II dose-finding studies. Br J Cancer. 2006 Mar 13;94(5):609-13. doi: 10.1038/sj.bjc.6602969. PMID 16434987
- [Derived] Herrera C, Lwanga J, Lee M, Mantori S, Amara A, Else L, Penchala SD, Egan D, Challenger E, Dickinson L, Boffito M, Shattock R, Khoo S, Fox J. Pharmacokinetic/pharmacodynamic investigation of raltegravir with or without lamivudine in the context of HIV-1 pre-exposure prophylaxis (PrEP). J Antimicrob Chemother. 2021 Jul 15;76(8):2129-2136. doi: 10.1093/jac/dkab136. PMID 33993302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were identified via study poster, internal recruitment emails, and via a list of individuals who had consented to be contacted for further research. Potential participants would contact the team, trial discussed & information sheet provided. If still interested, would be consented and screening visit booked.
Pre-assignment Details: Once participants were consented to the study, they undertook a screening visits to confirm eligibility. If eligibility was not confirmed, the participant was deemed a screen failure and not randomised to the trial.
Groups:
- Raltegravir, Then Raltegravir/Lamivudine: Raltegravir 400mg tablet, taken twice a day for 7days.
  Washout minimum of 28 days
  Raltegravir 400mg plus lamivudine 150mg taken twice a day for 7 days
- Raltegravir Lamivudine, Then Raltegravir: Raltegravir 400mg + Lamivudine 150mg tablet, taken twice a day for 7days.
  Washout minimum 28 days
  Raltegravir 400Mg Tab: bd for 7 days
Period: Phase 1
Arm/Group | Raltegravir, Then Raltegravir/Lamivudine | Raltegravir Lamivudine, Then Raltegravir
Started | 19 (One participant withdrawn and replaced. Data obtained from first participant still used in analysis) | 19 (One participant withdrawn and replaced. Data obtained from first participant still used in analysis)
Completed | 18 | 18
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1
Period: Phase 2
Arm/Group | Raltegravir, Then Raltegravir/Lamivudine | Raltegravir Lamivudine, Then Raltegravir
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Raltegravir, Then Raltegravir Plus Lamivudine: Raltegravir 400mg tablet, taken twice a day for 7days.
  Washout period 28 days
  Raltegravir 400mg + Lamivudine 150mg tablet, taken twice a day for 7days.
- Raltegravir Lamivudine, Then Raltegravir: Raltegravir 400mg + Lamivudine 150mg tablet, taken twice a day for 7days.
  Washout period 28 days
  Raltegravir 400Mg Tab: bd for 7 days
- Total: Total of all reporting groups
Arm/Group | Raltegravir, Then Raltegravir Plus Lamivudine | Raltegravir Lamivudine, Then Raltegravir | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (6.5) | 30.9 (8.0) | 29 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 16 | 10 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: The Level of Raltegravir Alone or Raltegravir /Lamivudine Required in the Plasma, Vagina and Rectum for 100% ex Vivo Protection From HIV
Description: The level of Raltegravir alone or Raltegravir /lamivudine required in the plasma, vagina and rectum for 100% ex vivo protection from HIV .
  High viral dose challenge: ex vivo challenge of tissue with 104 TCID50/mL HIV-1BaL Low viral dose challenge: ex vivo challenge of tissue with 102 TCID50/mL HIV-1BaL
Time Frame: Through Study completion, an average of 55 days
Population: Excludes two participants who were withdrawn from the study due to not meeting study inclusion criteria, but who were nonetheless included in safety analyses as they received at least one dose of study medication
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Raltegravir: Raltegravir 400mg tablet, taken twice a day for 7days.
  Raltegravir 400Mg Tab: bd for 7 days
- Raltegravir During Combination Treatment; Lamivudine During Combination Treatment: Raltegravir 400mg + Lamivudine 150mg tablet, taken twice a day for 7days.
  Raltegravir 400Mg Tab: bd for 7 days
  Lamivudine 150Mg Tablet: + Raltegravir 400Mg tablet bd for 7 days
Arm/Group | Raltegravir | Raltegravir During Combination Treatment | Lamivudine During Combination Treatment
Number analyzed (Participants) | 36 | 36 | 36
ng/mL
  Plasma: High Dose Challenge in rectal tissue | NA (NA) — Samples were below detection level for primary outcome | 669.90 (231.40) | 265.10 (76.50)
  Plasma: Low viral dose challenge in rectal tissue | 979.8 (306.5) | 669.90 (231.40) | 265.10 (76.50)
  Rectal: high viral dose challenge in rectal tissue | NA (NA) — Samples were below detection level for primary outcome | 862.35 (237.60) | 1722.02 (235.10)
  Rectal: Low viral dose challenge in rectal tissue | 729.36 (218.10) | 862.35 (237.60) | 1722.02 (235.10)
  Plasma: high viral dose challenge in vaginal tissu | NA (NA) — Samples were below detection level for primary outcome | 828.60 (510.30) | 266.40 (101.60)
  Plasma: low viral dose challenge in vaginal tissue | 979.8 (306.5) | 281.60 (99.10) | 169.10 (19.30)
  Plasma: high dose in vaginal tissue | NA (NA) — Samples were below detection level for primary outcome | 648.24 (432.90) | 1557.80 (206.30)
  Plasma: low dose in vaginal tissue | 607.60 (157.28) | 273.02 (88.40) | 1437.80 (133.30)

2. Secondary Outcome: The Time From First Dose of Drug to Maximum Mucosal ex Vivo Protection From HIV.
Description: Time in days from first receipt of antiretroviral (Raltegravir 400mg +/-lamivudine) until maximal ex vivo protection (against high or low titre of HIV-1BaL) was observed.
Time Frame: Up to 7 days from first dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Days
Groups:
- Raltegravir Lamivudine: Raltegravir 400mg + Lamivudine 150mg tablet, taken twice a day for 7days.
  Raltegravir 400Mg Tab: bd for 7 days
  Lamivudine 150Mg Tablet: + Raltegravir 400Mg tablet bd for 7 days
Arm/Group | Raltegravir | Raltegravir Lamivudine
Number analyzed (Participants) | 36 | 36
Days
  Time from first dose of drug to maximum rectal ex vivo protection from high titer HIV infection | 3 (0.58) | 2 (0)
  Time from first dose of drug to maximum rectal ex vivo protection from low titer HIV infection | 2 (0) | 2 (0)
  Time from first dose of drug to maximum rectal ex vivo protection from High titer HIV infection | 2.67 (0.67) | 3 (0.68)
  Time from first dose of drug to maximum vaginal ex vivo protection from low titer HIV infection | 3 (0.45) | 3.67 (0.61)

3. Secondary Outcome: Number of Adverse Events Based on PE, Blood Test and Event Reporting on Raltegravir Based PrEP, in HIV Negative Individuals
Description: Subject safety and tolerability will be determined by physical examination, blood tests and adverse event reporting. FBC, U&E and LFTs will be carried out at baseline and thereafter as symptom directed. Adverse event review. If significant adverse events have been reported, these will be clinically followed in accordance to the instruction of the study physician.
Time Frame: Through Study completion, an average of 55 days
Population: Includes two participants who were withdrawn from the study due to not meeting study inclusion criteria, but who were nonetheless included in safety analyses as they received at least one dose of study medication
Measure: Number; unit: Adverse event
Groups:
- Arm A Raltegravir: Raltegravir 400mg tablet, taken twice a day for 7days.
  Raltegravir 400Mg Tab: bd for 7 days
- Arm B Raltegravir Lamivudine: Raltegravir 400mg + Lamivudine 150mg tablet, taken twice a day for 7days.
  Raltegravir 400Mg Tab: bd for 7 days
  Lamivudine 150Mg Tablet: + Raltegravir 400Mg tablet bd for 7 days
Arm/Group | Arm A Raltegravir | Arm B Raltegravir Lamivudine
Number analyzed (Participants) | 38 | 38
Adverse event | 12 | 15

4. Secondary Outcome: The Time to Cessation of Mucosal ex Vivo Protection From HIV After Stopping ART at Steady State.
Description: Time in days from stopping antiretroviral (Raltegravir 400mg +/-lamivudine) until ex vivo protection (against high or low viral titre of HIV-1BaL) was no longer observed.
Time Frame: 5 days post last dose
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Days
Arm/Group | Raltegravir | Raltegravir Lamivudine
Number analyzed (Participants) | 36 | 36
Days
  Time to cessation of rectal ex vivo protection from high HIV dose challenge post ART at steady state | 3.33 (0.69) | NA (NA) — Cessation of mucosal ex vivo protection from HIV was not reached by the end of the follow up period (5 days), therefore mean and standard error could not be calculated.
  Time to cessation of rectal ex vivo protection from low HIV dose challenge post ART at steady state | NA (NA) — Cessation of mucosal ex vivo protection from HIV was not reached by the end of the follow up period (5 days), therefore mean and standard error could not be calculated. | NA (NA) — Cessation of mucosal ex vivo protection from HIV was not reached by the end of the follow up period (5 days), therefore mean and standard error could not be calculated.
  Time to cessation of vaginal ex vivo protection from high HIVdose challenge post ART at steady state | 4 (1.13) | NA (NA) — Cessation of mucosal ex vivo protection from HIV was not reached by the end of the follow up period (5 days), therefore mean and standard error could not be calculated.
  Time to cessation of vaginal ex vivo protection from low HIV dose challenge post ART at steady state | 5 (1.26) | NA (NA) — Cessation of mucosal ex vivo protection from HIV was not reached by the end of the follow up period (5 days), therefore mean and standard error could not be calculated.

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration each subject participated in the trial, this being from enrollment to final visit, which is approximately 55 days.
Description: All adverse event data that was captured as part of trial participation, including that of individuals withdrawn from the trial, were used in analysis
Arm/Group | Arm A Raltegravir | Arm B Raltegravir Lamivudine
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 12/38 | 15/38
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A Raltegravir (N=38) | Arm B Raltegravir Lamivudine (N=38)
Painful left toe (Musculoskeletal and connective tissue disorders) | 1 | 1
Viral illness with abdominal pain, vomiting, nausea, fever (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 1 | 3
Runny nose (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Abnormal LFTs (Blood and lymphatic system disorders) | 1 | 0
Acid Reflux (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Cold (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dehydration (General disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Dizziness (Nervous system disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
Fever (Infections and infestations) | 0 | 2
Flu (Infections and infestations) | 1 | 0
Fluoxetine Overdose (Injury, poisoning and procedural complications) | 0 | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Impacted tooth (Gastrointestinal disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Light headedness (Nervous system disorders) | 0 | 1
Loose Stool (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0
Neck lump right side (Blood and lymphatic system disorders) | 0 | 1
Nightmares and vivid dreams (Psychiatric disorders) | 0 | 5
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Perianal lump (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal Pain (General disorders) | 1 | 0
Rectal Discomfort and PR bleeding (Investigations) | 0 | 1
Sleep disturbance (Psychiatric disorders) | 0 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Spotting (Vascular disorders) | 0 | 2
Swollen neck glands (Blood and lymphatic system disorders) | 1 | 1
Tonsillitis (Infections and infestations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT03205566/Prot_SAP_000.pdf